CLINICAL TRIAL: NCT01029132
Title: Characteristics of Treatment Responders to Galantamine Administration in the Patients With Alzheimer's Disease
Brief Title: Characteristics of Treatment Responders to Galantamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Doh Kwan Kim, Principal Investigator, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-04-021
Record Dates: First submitted 2009-12-06; First posted 2009-12-09 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Dementia
Keywords: Alzheimer's disease; Galantamine; Treatment response; Efficacy; Adverse Event
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non-responder group (Experimental): patients who did not maintained or improved cognitive function
  Interventions: Drug: galantamine
- responder group (Experimental): patients who maintained or improved cognitive function
  Interventions: Drug: galantamine

INTERVENTIONS:
Drug: galantamine — 8 mg/day (4 mg bid) during the first 4 weeks, up to a maximum of 24 mg/day (12 mg bid) at intervals of 4 weeks, from 16 to 24 mg/day based on the patient's tolerability
  Other Names: galantamine-reminyl

SUMMARY:
To investigate the characteristics of treatment responders to galantamine.

DETAILED DESCRIPTION:
The purposes of this study are:

1. to investigate the characteristics of treatment responders to galantamine by examining the clinical response of galantamine in patients with mild to moderate AD for 52 weeks.
2. to examine the specific cognitive sub-domains that are more sensitive to galantamine administration.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of probable AD according to the criteria of the NINCDS-ADRDA
2. Korean version Mini-Mental State Examination scores between 10 and 26
3. History of cognitive decline that had been gradual in onset and progressive over at least 6 months
4. A caregiver who could assist the patient with medication, attend the assessment and provide information about the patient.

Exclusion Criteria:

1. they had evidence of any neurodegenerative diseases other than AD (i.e. Parkinson's disease, Huntington's disease)
2. Psychiatric disorder or severe behavioral disturbances that required psychotropic medications
3. Cerebral injuries induced by trauma, hypoxia, and/or ischemia
4. Clinically active cerebrovascular disease; History of seizure disorder
5. Other physical conditions that required acute treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale-preliminary Korean version (ADAS-cog-K) | baseline, 4w, 13w, 26w, 39w, 52w

SECONDARY OUTCOMES:
Seoul-Activities of Daily Living (S-ADL) Seoul-Instrumental Activities of Daily Living (S-IADL) Korean version Neuropsychiatric Inventory (K-NPI) | baseline, 4w, 13w, 26w, 39w, 52w

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, PhD, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea